CLINICAL TRIAL: NCT00216255
Title: An 8-week, Double-blind, Randomized, Multicenter, Flexible-dose, Placebo Controlled Pilot Study of Pagoclone in Patients With PDS Followed by a 52-week Open-label Extension
Brief Title: EXPRESS: Examining Pagoclone for Persistent Developmental Stuttering Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IP456-039
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Persistent Developmental Stuttering
Keywords: Persistent Developmental Stuttering
MeSH Terms: interventions — pagoclone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pagoclone (Experimental): .15mg, .30mg, .60mg
  Interventions: Drug: Pagoclone
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pagoclone
  Arms: Pagoclone
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of the study is to determine the effects of pagoclone on the symptoms of Persistent Developmental Stuttering, using a flexible dosing titration regimen on persistent developmental stuttering in patients 18 to 65 years of age.

ELIGIBILITY:
Inclusion Criteria:

* PDS defined as DSM-IV-TR criteria, symptoms starting before age 8, and a total overall score of 18-36 on the SSI-3
* English-speaking, with 8th grade education, able to understand and cooperate with study requirements without assistance
* Not pregnant or breastfeeding
* Able to consent

Exclusion Criteria:

* No diagnoses of other CNS/Mental health disorders in the last 6 months
* No use of psychotropic medication or other medication for stuttering within 4 weeks prior to screening
* No use of non-medicinal stuttering treatments for 5 months prior to the study
* No use of illicit drugs or opiates of any kind

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2005-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Effects of Pagaclone | 8 weeks double blind followed by a 52 weeks open label
  Primary objective using a flexible dosing titration regimen from 0.15mg Pagocolne BID, titrated at 2 weeks to 0.30mg Pagaclone BID for an additional 6 weeks versus placebo, on persistent developmental stuttering in patients 18 to 65 years of age over an 8 week, double blind treatment period, followed by five 53 week open label treatment extension periods. The primary efficacy variables will be based on data collected on the stuttering Severity Instrument-3 (SSI-3) Frequency and Duration Subscore, the Subjective Screening of Stuttering (SSS) Severity Subscore, and the treatment and week 8 visits. All efficacy assessments will evaluate change from pre-treatment to each on-treatment week.

SECONDARY OUTCOMES:
Secondary Objectives | Pre-treatment through week 8
  SSI-3 Total overall Score and individual subscores (including frequency, duration, and physical concomitant subscores) Subjective Screening of Stuttering (SSS) test Speech Naturalness Scales (SNS) Liebowitz Social Anxiety Scale (LSAS) Stuttering Clinician's Global Impression-Improvement (CGI) Optional Neuropsychological Test Optional Functional Brain Imaging

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Pivotal Research Centers, Peoria, Arizona
  - University of California, Irvine Medical School, Orange, California
  - Pharmacology Research Institute, Riverside, California
  - Pacific Clinical Research Medical Group, Upland, California
  - University of South Florida College of Medicine, Tampa, Florida
  - Atlanta Institute of Medicine & Research-Atlanta Clinic, Atlanta, Georgia
  - Davis Clinic PC, Indianapolis, Indiana
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Pivotal Research Centers, Royal Oak, Michigan
  - Social Psychiatry Research Institute, Brooklyn, New York
  - Social Psychiatry Research Institute, New York, New York
  - Midwest Clinical Research Center, Dayton, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - FutureSearch Trials, Austin, Texas
  - University of Texas, Health Science Center, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- See also: Related Info — http://www.stutteringstudy.com